CLINICAL TRIAL: NCT02149277
Title: Effects of Exogenous Recombinant GCSF in Patients With Repeated Implantation Failure - A Randomized Single-blind Trial
Brief Title: Gcsf Injection in Women With Repeated Implantaiton Failure
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment difficulty
Sponsor: Clinique Ovo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ovo-12-06
Record Dates: First submitted 2014-03-19; First posted 2014-05-29 (Estimated); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Repeated Embryo Implantation Failure
Keywords: Infertility; IVF; Embryo transfer
MeSH Terms: conditions — Infertility | interventions — Filgrastim

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Filgrastim (Active Comparator): Injection Filgrastim 300 ug intravaginally during an IVF cycle or during an embryo transfer
  Interventions: Drug: Filgrastim
- Sodium Chloride (Placebo Comparator): Injection of 1 ml of Sodium Chloride intravaginally during an IVF cycle or during an embryo transfer cycle.
  Interventions: Drug: Filgrastim

INTERVENTIONS:
Drug: Filgrastim — The fertility specialist will inject the study medication or its placebo on the 6th day of gonadotrophin stimulation for IVF subjects. For the subjects undergoing embryo transfer, the injection will be done once the endometrial lining measure more than 8mm.
  Other Names: Neupogen

SUMMARY:
The purpose of the study is to see the impact of intrauterine injection of recombinant GCSF on pregnancy and implantation rate during IVF-ICSI (intracytoplasmic sperm injection) protocols as well as in frozen embryo transfer. In addition, following the injection, the level of G-CSF in the bloodstream will be verified.

DETAILED DESCRIPTION:
Recently, scientists have been interested in G-CSF (Granulocyte - Colony Stimulating Factor) and the latter has seen its use grow in reproductive pathology.

G -CSF, a true center pivot, would act concurrently on oocyte quality and endometrial receptivity, improving:

* Immune tolerance
* The self-healing of oocyte chromosome abnormalities
* The adherence of the embryo

The injection of G-CSF molecule has been used in different circumstances. One of its uses, among others, is to help rebuild the immune system in patients undergoing chemotherapy. Some studies have been conducted in patients having embryo implantation problems; they have demonstrated improved rates of pregnancy and childbirth after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18 and 37
* Indication of the Antagonist IVF protocol or indication of a substituted frozen embryo transfer
* Subjects with repetitive embryo implantation failure meaning: a history of 3 embryos transferred including frozen embryo without a positive pregnancy test for women 35 years and younger
* Subjects with repetitive embryo implantation failure meaning: a history of 4 embryos transferred including frozen embryo without a positive pregnancy test for women between the ages of 35 and 37.
* Negative repetitive implantation failure work up

Exclusion Criteria:

* Renal failure or cardiac failure
* Chronic neutropenia
* Past or present cancer history
* Sickle cell anemia
* Lithium treatment
* Voluntary withdrawal from the study
* Use of concomitant medication: DHEA (dehydroepiandrosterone ), CoQ10 (coenzyme Q10), Growth Hormone and Viagra

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Dosage of G-CSF | up to 3 years
  Measure dosage of G-CSF in the bloodstream on the day of oocyte retrieval and measure the implantation rate as well as pregnancy rate following the G-CSF injection
Pregnancy and Implantation | up to 3 years
  Measure the pregnancy and embryo implantation rate post G-CSF injection

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Kadoch, Md, Principal Investigator — Clinique Ovo
Locations (1):
- Clinique Ovo, Montreal, Quebec, Canada